CLINICAL TRIAL: NCT02772822
Title: A Phase Ⅲ, Multi-center, Randomized, Controlled Study to Compare the Efficiency and Safety of SCT400(Recombinant Chimeric Anti-CD20 Monoclonal Antibody, Experimental Drug) Plus CHOP Versus Rituximab Plus CHOP in Untreated CD20-positive DLBCL Patients
Brief Title: A Study Comparing the Efficiency and Safety of S-CHOP(Cyclophosphamide, Hydroxydaunomycin, Oncovin, and Prednisone) Versus R-CHOP in Untreated CD20(Cluster of Differentiation Antigen 20)-Positive DLBCL Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCT400NHL3
Record Dates: First submitted 2016-05-06; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): SCT400 plus CHOP, six cycles SCT400: 375 mg/m2, IV, day 1 of each cycle Cyclophosphamide: 750 mg/m2, IV, day 2 of each cycle Doxorubicin: 50 mg/m2, IV, day 2 of each cycle Vincristine: 1.4 mg/m2, up to a maximal dose of 2 mg, IV, day 2 of each cycle Prednisone: 100 mg, po, day 2 to day 6 of each cycle
  Interventions: Drug: SCT400 plus CHOP
- Active Comparator (Active Comparator): Rituximab plus CHOP, six cycles Rituximab: 375 mg/m2, IV, day 1 of each cycle Cyclophosphamide: 750 mg/m2, IV, day 2 of each cycle Doxorubicin: 50 mg/m2, IV, day 2 of each cycle Vincristine: 1.4 mg/m2, up to a maximal dose of 2 mg, IV, day 2 of each cycle Prednisone: 100 mg, po, day 2 to day 6 of each cycle
  Interventions: Drug: Rituximab plus CHOP

INTERVENTIONS:
Drug: SCT400 plus CHOP
  Arms: Experimental
Drug: Rituximab plus CHOP
  Arms: Active Comparator

SUMMARY:
The primary objective of the study is to assess the efficiency of SCT400 plus CHOP versus Rituximab plus CHOP in untreated CD20-positive DLBCL Patients.

The secondary objective of the study is to evaluate the safety of SCT400 plus CHOP, as well as the presence of human anti-chimeric antibodies (HACA).

ELIGIBILITY:
Inclusion Criteria:

1. Untreated CD20-positive DLBCL confirmed by local histopathology.
2. International Prognostic Index (IPI) score of 0 to 2:

   Score 0 needs to accompanied by bulky disease, which is defined as the presence of a tumor mass with a diameter of more than 7.5 cm.
3. 18 years to 70 years; Male or female patients.
4. More than 6 months life expectancy.
5. At least one measurable lymph node:

   For nodal tumor mass, more than 1.5 cm in the long axis and more than 1.0 cm in the short axis; For extranodal tumor mass, more than 1.0 cm in the long axis.
6. Eastern Cooperative Oncology Group(ECOG) performance status of 0 to 2.
7. Adequate cardiac function (LVEF≥50%).
8. Adequate hematological function: absolute neutrophil count(ANC) ≥1.5*109/L and platelet count(PLT) ≥75*109/L.
9. Fertile patients must use effective contraception during the treatment and within 3 months after the treatment.
10. Signed an informed consent form which was approved by the institutional review board of the respective medical center.

Exclusion Criteria:

1. Known allergic reactions against human or murine monoclonal antibody, murine products, or foreign proteins.
2. Known allergic reactions against any component of CHOP regimen.
3. Previous treatment for DLBCL, including chemotherapy, immunotherapy, partial radiotherapy for lymphoma, monoclonal antibody therapy or surgical treatment (excluding lymph node biopsies and surgical resection for non-lymphoma lesions).
4. History of cytotoxic drugs treatment or anti-CD20 monoclonal antibody treatment for other disease (e.g., rheumatoid arthritis), or prior use of any monoclonal antibody within 3 months.
5. Primary central nervous system(CNS) lymphoma, secondary CNS involvement, grey zone lymphoma (GZL) between burkitt and DLBCL, primary effusion lymphoma, plasmablastic lymphoma, primary cutaneous DLBCL, anaplastic lymphoma kinase(ALK) positive DLBCL or transformed lymphoma.
6. History of other cancer within the past 5 years except cured basal cell skin cancer, squamous cell carcinoma, cutaneous melanoma or carcinoma in situ of the cervix.
7. Patients who have significant cardiac disease, including heart disease of grade Ⅲ of Ⅳ according to the New York Heart Association(NYHA) system, or occurrence of myocardial infarction, unstable arrhythmia, unstable angina or severe hypertension in the past 6 months or peripheral nervous system(PNS) or CNS disease.
8. Previously suffered from progressive multifocal leukoencephalopathy.
9. Having continuous treatment of corticosteroid drugs lasting for more than 10 days:

   Prednisone with the dosage over 30mg/day; Other corticosteroid drugs with equal dosage.
10. Participation in another clinical trial in the past 3 months.
11. Recent major surgery within 4 weeks.
12. Use of hemopoietic cytokine in the past 2 weeks, e.g. granulocyte colony stimulating factor(G-CSF).
13. Vaccination with a attenuated live vaccine within 4 weeks.
14. Abnormal laboratory values:

    Creatinine more than 1.5 times normal value; Aspartate aminotransferase(AST) or alanine aminotransferase(ALT) more than 2.5 times normal value (5 times if hepatic involvement); total bilirubin(T-BIT) more than 1.5 times normal value(3 times if hepatic involvement); Without anticoagulant therapy, partial thromboplastin time(PTT), activated partial thromboplastin time(APTT) or international normalized ratio(INR) more than 1.5 times normal value.
15. Active Infectious disease or significant infections requiring intravenous antibiotic therapy or hospitalization in the past 4 weeks (exception of tumor induced fever).
16. Suspected active or latent tuberculosis.
17. Seropositive for human immunodeficiency virus (HIV) or hepatitis C antibodies. Hepatitis B virus(HBV) positive patient (including positive hepatitis B surface antigen or positive hepatitis B virus core antibody) may participate if his serum HBV DNA level is sufficient low.
18. Other disease or symptom by the investigator's discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) after completion of treatment | 18 weeks

SECONDARY OUTCOMES:
Complete remission(CR) plus complete remission/unconfirmed(CRu) after completion of treatment | 18 weeks
Progression-free survival(PFS) | 1 year
Event-free survival(EFS) at 1 year and directly after an event, whichever comes first. The events are defined as progressive disease, relapse, death from any cause, or new anticancer treatment | 1 year
Duration of remission(DOR) measured from prior achievement of complete remission or partial remission to occurrence of an event or at 1 year, whichever comes first. The events are defined as progressive disease, relapse of death from any cause | 1 year
Overall survival(OS) | 1 year
Comparison of adverse events(AEs) between the two study arms | 1 year
Number of participants with seropositive for human anti-chimeric antibody(HACA) between the two study arms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yuan kai Shi, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Beijing， China
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No